CLINICAL TRIAL: NCT04204642
Title: SEarchiNg BiomarkErs Cerebral Amyloid Angiopathy (SENECA): Italian Network for the Study of CAA
Brief Title: SEarchiNg BiomarkErs Cerebral Amyloid Angiopathy (SENECA)
Acronym: SENECA
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: SENECA
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Amyloid Angiopathy
MeSH Terms: conditions — Cerebral Amyloid Angiopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A peripheral blood withdrawal for APOE allele screening will be performed in all patients, after informed consent obtainment. Additionally, cases with early onset clinical manifestations and/or rapid clinical progression and/or relatives with a diagnosis of CAA or presenting early onset CAA clinical features will be addressed to the genetic screening of Amyloid Precursor Protein (APP) and Transthyretin (TTR) gene. A subgroup of patients will undergo at T0, T1 and T2 a whole venous blood withdrawal, to collect serum and plasma samples, evaluate the platelet concentration of Aβ40 by thioflavin T (ThT) assay and Western blot analysis and the inflammatory and endothelial profile of CAA patients by ELISA or Bio-Plex Panels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cerebral amyloid angiopathy (CAA): Cerebral amyloid angiopathy (CAA) patients
  Interventions: Other: CAA patients data collection

INTERVENTIONS:
Other: CAA patients data collection — Demographic and clinical data of each patient, including index event that led to the diagnosis (cerebrovascular disease, dementia, gait disturbance, TFNE, seizures, headache), vascular risk factors, history of brain injury or neurosurgery, familial history, and pharmacological treatment will be collected by neurologists in charge.
  Other Names: Prognostic factors evaluation

SUMMARY:
Cerebral amyloid angiopathy (CAA) is one of the major types of cerebral small vessel disease, and a leading cause of spontaneous intracerebral hemorrhage and cognitive decline in elderly patients. Although increasingly detected, a number of aspects including the pathophysiology, the clinical and neuroradiological phenotype and the disease course are still under investigation. The incomplete knowledge of the disease limits the implementation of evidence based guidelines on patient's clinical management and the development of treatments able to prevent or reduce disease progression.

The SENECA (SEarchiNg biomarkErs of Cerebral Angiopathy) project is the first Italian multicentre cohort study aimed at better defining the disease natural history and identifying clinical and neuroradiological markers of disease progression. By a multidisciplinary approach and the collection of a large and well phenotyped series and biorepository of CAA patients, the study is ultimately expected to improve the diagnosis and the knowledge of CAA pathophysiological mechanisms.

DETAILED DESCRIPTION:
The SENECA is an Italian multicenter network integrating the experience of neurologists, neuroradiologists, neuro-ophthalmologists and biologists and allowing the standardized collection of a well-characterized wide series of sporadic and familial CAA patients.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients ≥55 years (with the exception of genetic cases), referred to the participating centres, with a diagnosis of possible probable and definite symptomatic or asymptomatic CAA, defined according to the modified Boston neuroradiological criteria, who had undergone at least one brain MRI (mandatory requirement for inclusion of the patient in the study) will be recruited.

Exclusion Criteria:

* evidence of other causes of cerebral hemorrhage (brain tumors, arteriovenous malformations, aneurysms, cavernous angiomas), contraindications to brain MRI, pregnancy and breastfeeding

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sporadic and familial CAA patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical and neuroradiological phenotype | 24 months
  description of the phenotypic characteristics of a large population of CAA patients collected in Italy

SECONDARY OUTCOMES:
severity of the neuroradiological picture | 24 months
  Evaluation of the severity of the neuroradiological picture (presence and site of WMHs, CMBs, cSS, CMIs, EPVS ,global cortical atrophy and SAH)

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Neurologia 5, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Storti B, Marinoni G, Cefaloni B, Francia A, Rifino N, Boncoraglio G, Indaco A, Di Fede G, Stanziano M, Canavero I, Bersano A. Cerebrospinal Fluid Biomarkers in Cerebral Amyloid Angiopathy With and Without Spontaneous Lobar Hemorrhage. J Am Heart Assoc. 2025 Sep 16;14(18):e042445. doi: 10.1161/JAHA.125.042445. Epub 2025 Sep 11. PMID 40932118
- [Derived] Storti B, Stanziano M, Marinoni G, Mazze A, Francia A, Zacarias E, Strazzabosco C, De Toma C, Rifino N, Boncoraglio G, Di Fede G, Pollaci G, Gatti L, Canavero I, Bersano A. Hippocampal Subfields Volume: Another Hint of the Continuum Between CAA and AD? Eur J Neurol. 2025 Jul;32(7):e70284. doi: 10.1111/ene.70284. PMID 40626372